CLINICAL TRIAL: NCT02178475
Title: Prospective Observational Study of Febrile Neutropenia (FN) and Pegfilgrastim Primary Prophylaxis in Breast Cancer and Non-Hodgkin's Lymphoma Patients Receiving High (>20%) FN-risk Chemotherapy
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120214
Record Dates: First submitted 2014-06-10; First posted 2014-06-30 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-10

CONDITIONS: Chemotherapy-induced Febrile Neutropenia
Keywords: NHL; Breast Cancer
MeSH Terms: conditions — Chemotherapy-Induced Febrile Neutropenia; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chemotherapy + Pegfilgrastim: Patients with non-Hodgkin's lymphoma or breast cancer being treated with a permitted standard-dose chemotherapy regimen with a high FN risk (> 20%) and who had pegfilgrastim prophylaxis initiated in the first cycle of chemotherapy.

SUMMARY:
To estimate the incidence of febrile neutropenia in patients with breast cancer and non-Hodgkin's lymphoma receiving high (> 20%) FN-risk chemotherapy and pegfilgrastim primary prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Any stage NHL or breast cancer and received the first cycle of a new chemotherapy course.
* Received the first cycle of a permitted standard dose chemotherapy regimens with an estimated high (> 20%) FN risk according to published data or guidelines (dose modifications +/-10% in Cycle 1 are allowable).
* Initiated treatment in Cycle 1 with pegfilgrastim according to the pegfilgrastim summary of product characteristics. (SmPC). Enrolment must occur after the first pegfilgrastim dosing in Cycle 1 and before the second day of Cycle 2.

Exclusion Criteria:

* Ongoing or planned concurrent participation in any clinical study involving Investigational Product that has not been approved by the national competent authorities for any indication.
* Ongoing or planned concurrent participation in any clinical study where the administration of Colony Stimulating Factor (CSF) is determined by the protocol (clinical trials on an approved drug and observational trials are permitted as long as these do not mandate how neutropenia should be treated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NHL or breast cancer who have initiated treatment with a permitted standard-dose chemotherapy regimen that has a high FN risk (> 20%) per published studies or international guidelines, and who started pegfilgrastim in Cycle 1
Sampling Method: Probability Sample
Enrollment: 943 (Actual)
Dates: Start 2014-07-18 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (60):
- Austria (5):
  - Research Site, Eggenburg
  - Research Site, Graz
  - Research Site, Leoben
  - Research Site, Schwarzach im Pongau
  - Research Site, Vienna
- Belgium (2):
  - Research Site, Arlon
  - Research Site, Liège
- Bulgaria (2):
  - Research Site, Pleven
  - Research Site, Sofia
- Czechia (5):
  - Research Site, Chomutov
  - Research Site, Hořovice
  - Research Site, Nový Jičín
  - Research Site, Pilsen
  - Research Site, Prague
- France (14):
  - Research Site, Aix-en-Provence
  - Research Site, Amiens
  - Research Site, Beuvry
  - Research Site, Marseille
  - Research Site, Meaux
  - Research Site, Nancy
  - Research Site, Nîmes
  - Research Site, Orléans
  - Research Site, Perpignan
  - Research Site, Périgueux
  - Research Site, Pierre-Bénite
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Sarcelles
  - Research Site, Strasbourg
- Germany (9):
  - Research Site, Bonn
  - Research Site, Dresden
  - Research Site, Fulda
  - Research Site, Hildesheim
  - Research Site, Kassel
  - Research Site, Stolberg
  - Research Site, Troisdorf
  - Research Site, Velbert
  - Research Site, Westerstede
- Greece (8):
  - Research Site, Athens
  - Research Site, Chania
  - Research Site, Kalamata
  - Research Site, Larissa
  - Research Site, Nea Kifissia, Athens
  - Research Site, Papagou
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gdynia
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wałbrzych
- Romania (8):
  - Research Site, Baia Mare
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Câmpina
  - Research Site, Cluj-Napoca
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Ploieşti

REFERENCES:
- [Derived] Mahtani RL, Belani R, Crawford J, Dale D, DeCosta L, Gawade PL, Huynh C, Lawrence T, Lewis S, MacLaughlin WW, Narang M, Rifkin R. A prospective cohort study to evaluate the incidence of febrile neutropenia in patients receiving pegfilgrastim on-body injector versus other options for prophylaxis of febrile neutropenia: breast cancer subgroup analysis. Support Care Cancer. 2022 Jul;30(7):6135-6144. doi: 10.1007/s00520-022-07025-2. Epub 2022 Apr 14. PMID 35426046
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 66 centers in Austria, Belgium, Bulgaria, Czech Republic, France, Germany, Greece, Poland, and Romania. The first participant enrolled on 18 July 2014 and the last participant enrolled on 28 April 2016.
Pre-assignment Details: Participants were enrolled at sites where they were receiving treatment as part of their routine standard of care. No specific interventional tests, investigations, procedures or changes to routine practice were conducted as part of this study.
Period: Overall Study
Arm/Group | Chemotherapy + Pegfilgrastim
Started | 943
Primary Analysis Set | 844 (All enrolled participants who met eligibility criteria)
Completed | 814
Not Completed | 129
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 10
Not completed — Death | 13
Not completed — Protocol-specified Criteria | 99

BASELINE CHARACTERISTICS:
Population: Primary Analysis Set
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 844
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.2)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 563
  ≥ 65 years | 281
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 723
  Male | 121
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 4
  White | 673
  Other | 1
  Missing | 166
Tumor Type [Count of Participants; unit: Participants]
  Non-Hodgkin's lymphoma (NHL) | 190
  Breast cancer | 654
Baseline Comorbidities [Number; unit: participants] — COPD = chronic obstructive pulmonary disease
  participants
    Liver disease | 18
    Cardiovascular disease | 211
    Diabetes mellitus | 75
    COPD/Pulmonary disease | 41
    Renal disease/impaired clearance | 16
    Current infection | 8
    Open wound | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 645
    1 (Restrictive but ambulatory) | 129
    2 (Ambulatory but unable to work) | 14
    3 (Limited self-care) | 6
    4 (Disabled, confined to bed/chair) | 1
    Missing | 49
History of Febrile Neutropenia [Count of Participants; unit: Participants]
  Yes | 5
  No | 839

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Febrile Neutropenia
Description: Febrile neutropenia (FN) was defined as an absolute neutrophil count (ANC) of < 0.5 x 10^9/L, or < 1.0 x 10^9/L predicted to fall below 0.5 x 10^9/L within 48 hours with fever or clinical signs of sepsis; fever and ANC were measured the same day or within ± 1 calendar day.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 844
percentage of participants
  Overall | 3.3 [2.3 to 4.8]
  Cycle 1 | 1.9 [1.2 to 3.1]
  Cycle 2: number analyzed (Participants) | 824
  Cycle 2 | 0.4 [0.1 to 1.1]
  Cycle 3: number analyzed (Participants) | 803
  Cycle 3 | 0.5 [0.2 to 1.3]
  Cycle 4: number analyzed (Participants) | 760
  Cycle 4 | 0.5 [0.2 to 1.3]
  Cycle 5: number analyzed (Participants) | 694
  Cycle 5 | 0.3 [0.1 to 1.0]
  Cycle 6: number analyzed (Participants) | 666
  Cycle 6 | 0.3 [0.1 to 1.1]
  Cycle 7: number analyzed (Participants) | 232
  Cycle 7 | 0.0 [0.0 to 1.6]
  Cycle 8: number analyzed (Participants) | 226
  Cycle 8 | 0.0 [0.0 to 1.7]

2. Secondary Outcome: Number of Participants Who Discontinued Pegfilgrastim Prophylaxis
Description: Participants who discontinued pegfilgrastim prophylaxis was defined as participants who received at least one cycle of chemotherapy (cycle 2 or later) in which pegfilgrastim prophylaxis was not administered, but other granulocyte colony-stimulating factor (G-CSF) prophylaxis was administered. Participants in this group received either pegfilgrastim or other G-CSF prophylaxis in all chemotherapy cycles.
  Discontinuation was categorized as either temporary (participant received pegfilgrastim prophylaxis in at least one subsequent cycle) or permanent (participant had at least one cycle of chemotherapy following the cycle in which no pegfilgrastim prophylaxis was administered, and other G-CSF prophylaxis (i.e. not pegfilgrastim) was administered in all subsequent cycles, OR participant did not receive pegfilgrastim prophylaxis in the last cycle of chemotherapy, and other G-CSF prophylaxis was administered).
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Primary analysis set
Measure: Number; unit: participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 844
participants
  Discontinuation of pegfilgrastim prophylaxis | 26
  Temporary discontinuation | 4
  Permanent discontinuation | 22

3. Secondary Outcome: Number of Participants Who Discontinued G-CSF Prophylaxis
Description: Participants who discontinued G-CSF prophylaxis was defined as participants who received at least one cycle of chemotherapy (cycle 2 or later) in which no G-CSF prophylaxis was administered.
  Discontinuation was categorized as either temporary (participant received G-CSF prophylaxis in at least one subsequent cycle) or permanent (participant had at least one cycle of chemotherapy following the cycle in which no G-CSF prophylaxis was administered, and no G-CSF prophylaxis was administered in any subsequent cycle, OR participant did not receive G-CSF prophylaxis in the last cycle of chemotherapy).
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Primary analysis set
Measure: Number; unit: participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 844
participants
  Discontinuation of G-CSF prophylaxis | 44
  Temporary discontinuation | 9
  Permanent discontinuation | 35

4. Secondary Outcome: Characteristics of Participants Who Discontinued Pegfilgrastim Prophylaxis
Description: Participants who discontinued pegfilgrastim prophylaxis are participants who received at least one cycle of chemotherapy (cycle 2 or later) in which pegfilgrastim prophylaxis was not administered, but other G-CSF prophylaxis was administered in this cycle. Participants in this group received either pegfilgrastim or other G-CSF prophylaxis in all chemotherapy cycles.
  Data includes both temporary and permanent pegfilgrastim discontinuation.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Participants who received at least 1 cycle of chemotherapy in which no pegfilgrastim prophylaxis was administered, but another G-CSF was administered.
Measure: Number; unit: participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 26
participants
  Male | 6
  Female | 20
  Race: Black | 0
  Race: White | 15
  Race: Missing | 11
  Age < 65 years | 15
  Age ≥ 65 years | 11
  Age ≥ 75 years | 1
  Tumor type: NHL | 15
  Tumor type: Breast cancer | 11

5. Secondary Outcome: Characteristics of Participants Who Discontinued G-CSF Prophylaxis
Description: Participants who discontinued G-CSF prophylaxis are participants who received at least one cycle of chemotherapy (cycle 2 or later) in which no G-CSF prophylaxis was administered.
  Data includes both temporary and permanent discontinuation of G-CSF prophylaxis.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Participants who received at least 1 cycle of chemotherapy in which no G-CSF prophylaxis was administered.
Measure: Number; unit: participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 44
participants
  Male | 8
  Female | 36
  Race: Black | 0
  Race: White | 36
  Race: Missing | 8
  Age < 65 years | 26
  Age ≥ 65 years | 18
  Age ≥ 75 years | 2
  Tumor type: NHL | 13
  Tumor type: Breast cancer | 31

6. Secondary Outcome: Number of Cycles With No Pegfilgrastim Prophylaxis
Description: A cycle of chemotherapy (cycle 2 or later) in which pegfilgrastim prophylaxis was not administered, but other G-CSF prophylaxis was administered in this cycle.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: All cycles of chemotherapy for participants in the primary analysis set
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 844
Number analyzed (cycles) | 5049
cycles | 56

7. Secondary Outcome: Number of Cycles With no G-CSF Prophylaxis
Description: A cycle of chemotherapy (cycle 2 or later) in which no G-CSF prophylaxis was administered.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: All cycles of chemotherapy for participants in the primary analysis set
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 844
Number analyzed (cycles) | 5049
cycles | 105

8. Secondary Outcome: Reasons for Discontinuation of Pegfilgrastim Prophylaxis
Description: as for outcome 4
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 26
Participants
  Daily G-CSF preferred to once-per-cycle G-CSF | 14
  Cost | 1
  Following protocol of hospital or country/region | 2
  Adverse reaction to G-CSF | 6
  Other | 3

9. Secondary Outcome: Reasons for Discontinuation of G-CSF Prophylaxis
Description: Participants who discontinued G-CSF prophylaxis are participants who received at least one cycle of chemotherapy (cycle 2 or later) in which no G-CSF prophylaxis was administered.
  Data includes both temporary and permanent discontinuation of G-CSF prophylaxis. Participants may have more than 1 discontinuation reason.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Participants who received at least 1 cycle of chemotherapy in which no G-CSF prophylaxis was administered.
Measure: Number; unit: participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 44
participants
  Chemotherapy dose intensity reduced | 9
  Patient no longer considered at high risk of FN | 14
  Cost | 3
  Following protocol of hospital or country/region | 2
  Adverse reaction to G-CSF | 3
  Other | 22
  Missing | 2

10. Secondary Outcome: Percentage of Participants Who Experienced Complications of Febrile Neutropenia
Description: Complications of febrile neutropenia were defined as FN-related hospitalizations and death, and neutropenia-related chemotherapy dose delays and dose reductions.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 844
percentage of participants | 6.8 [5.2 to 8.7]

11. Secondary Outcome: Number of Febrile Neutropenia Events That Occurred During Cycles With No G-CSF Prophylaxis
Description: The number of febrile neutropenia events that occurred during a cycle of chemotherapy (cycle 2 or later) in which no G-CSF prophylaxis was administered. Febrile neutropenia was defined as an ANC of < 0.5 x 10^9/L, or < 1.0 x 10^9/L predicted to fall below 0.5 x 10^9/L within 48 hours with fever or clinical signs of sepsis; fever and ANC were measured the same day or within ± 1 calendar day.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: All FN events observed for participants in the primary analysis set
Measure: Number; unit: febrile neutropenia events
Units Other Than Participants: febrile neutropenia events
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 844
Number analyzed (febrile neutropenia events) | 31
febrile neutropenia events | 2

12. Secondary Outcome: Number of Participants Who Experienced Febrile Neutropenia During Cycles With No G-CSF Prophylaxis
Description: The number of participants who received at least one cycle of chemotherapy in which no G-CSF prophylaxis was administered who experienced febrile neutropenia during a cycle of chemotherapy in which no G-CSF prophylaxis was administered. Febrile neutropenia was defined as an ANC of < 0.5 x 10^9/L, or < 1.0 x 10^9/L predicted to fall below 0.5 x 10^9/L within 48 hours with fever or clinical signs of sepsis; fever and ANC were measured the same day or within ± 1 calendar day.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Participants who received at least 1 cycle of chemotherapy in which no G-CSF prophylaxis was administered.
Measure: Number; unit: participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 44
participants | 2

13. Secondary Outcome: Number of Participants Who Experienced Complications of Febrile Neutropenia During Cycles With No G-CSF Prophylaxis
Description: The number of participants who received at least one cycle of chemotherapy in which no G-CSF prophylaxis was administered who experienced complications of febrile neutropenia during a cycle of chemotherapy in which no G-CSF prophylaxis was administered. Complications of febrile neutropenia were defined as FN-related hospitalizations and death, and neutropenia-related chemotherapy dose delays and dose reductions.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Participants who received at least 1 cycle of chemotherapy in which no G-CSF prophylaxis was administered
Measure: Number; unit: participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 44
participants | 3

14. Secondary Outcome: Number of Cycles With No G-CSF Prophylaxis in Which Febrile Neutropenia Events Occurred
Description: The number of chemotherapy cycles during which an event of febrile neutropenia occurred in which no G-CSF prophylaxis was administered. Febrile neutropenia was defined as an ANC of < 0.5 x 10^9/L, or < 1.0 x 10^9/L predicted to fall below 0.5 x 10^9/L within 48 hours with fever or clinical signs of sepsis; fever and ANC were measured the same day or within ± 1 calendar day.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Cycles of chemotherapy for participants who received at least one cycle of chemotherapy in which no G-CSF prophylaxis was administered.
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 44
Number analyzed (cycles) | 105
cycles | 2

15. Secondary Outcome: Number of Cycles With No G-CSF Prophylaxis in Which Complications of Febrile Neutropenia Occurred
Description: The number of chemotherapy cycles during which complications of febrile neutropenia occurred in which no G-CSF prophylaxis was administered. Complications of febrile neutropenia were defined as FN-related hospitalizations and death, and neutropenia-related chemotherapy dose delays and dose reductions.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Cycles of chemotherapy for participants who received at least one cycle of chemotherapy in which no G-CSF prophylaxis was administered, in which no G-CSF prophylaxis was administered.
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 44
Number analyzed (cycles) | 105
cycles | 3

16. Secondary Outcome: Number of Participants Who Permanently Switched From Pegfilgrastim Prophylaxis to Other G-CSF Prophylaxis
Description: The number of participants who received pegfilgrastim prophylaxis from cycle 1 until a cycle when other G-CSF prophylaxis was administered, and this G-CSF or a different G-CSF agent (not pegfilgrastim) was received as prophylaxis at each remaining cycle of the chemotherapy course.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Primary analysis set
Measure: Number; unit: participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 844
participants | 22

17. Secondary Outcome: Characteristics of Participants Who Received On-schedule Pegfilgrastim Primary Prophylaxis
Description: On-schedule pegfilgrastim primary prophylaxis was defined as participants who received pegfilgrastim in cycle 1 and continued to receive pegfilgrastim across all cycles, administered 1-3 days after the end of cytotoxic chemotherapy in each cycle.
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Population: Participants who received pegfilgrastim across all cycles, administered 1- 3 days after the end of cytotoxic chemotherapy in each cycle.
Measure: Number; unit: participants
Arm/Group | Chemotherapy + Pegfilgrastim
Number analyzed (Participants) | 683
participants
  Male | 72
  Female | 611
  Race: White | 546
  Race: Black or African American | 2
  Race: Other | 1
  Race: Missing | 134
  Age < 65 years | 464
  Age ≥ 65 years | 219
  Age ≥ 75 years | 38
  Tumor type: NHL | 112
  Tumor type: Breast cancer | 571

ADVERSE EVENTS:
Time Frame: Participants were followed for up to 8 cycles of chemotherapy; the average observation time was 4.1 months.
Description: In this observational study only adverse events deemed to be related to study drug (adverse drug reactions; ADRs) were collected.
  Other Adverse Events summarizes the non-serious occurrences of ADRs that exceed the indicated frequency threshold.
Arm/Group | Chemotherapy + Pegfilgrastim
Serious Adverse Events (participants affected / at risk) | 5/844
Other Adverse Events (participants affected / at risk) | 11/844
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Pegfilgrastim (N=844)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Pegfilgrastim (N=844)
Bone pain (Musculoskeletal and connective tissue disorders) | 11

LIMITATIONS AND CAVEATS:
The study had planned to enroll equal numbers of subjects with NHL and breast cancer; however, more patients with breast cancer were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.